CLINICAL TRIAL: NCT06853548
Title: Investigation of the Relationship Between Core Stability and Respiratory Parameters in Children With Thoracic Hyperkyphosis
Brief Title: Core Stability and Respiratory Parameters in Children With Thoracic Hyperkyphosis
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Kubra Koce, Lecturer, Istinye University
Other Study IDs: 24-02
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Hyperkyphosis; Respiratory Failure
Keywords: Thoracic Hyperkyphosis; Respiratory Function; Respiratory Muscle Strength; Core Stability
MeSH Terms: conditions — Kyphosis; Respiratory Insufficiency; Respiratory Aspiration | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment — Respiratory function, respiratory muscle strength, and core stability parameters will be assessed in children with hyperkyphosis.

SUMMARY:
Hyperkyphosis, defined as an excessive curvature of the thoracic spine beyond normal limits, is among the factors that reduce chest wall mobility and lung function. In modern society, increased sitting durations contribute to increased thoracic kyphosis. Studies have indicated that an increase in thoracic kyphosis and a decrease in thoracic spinal mobility are associated with reduced respiratory functions, such as forced vital capacity (FVC) and forced expiratory volume in one second (FEV1).

The diaphragm forms the upper part of the core stability system. When contracted, it increases intra-abdominal pressure, contributing to core stability. The diaphragm also contracts in advance of and during limb movements to assist in postural control. Additionally, the diaphragm is the primary respiratory muscle responsible for inspiration. Any functional loss in the diaphragm, which alone accounts for 65-80% of vital capacity, can significantly reduce inspiratory capacity. During forced expiration, muscles such as the rectus abdominis, transversus abdominis, internal obliques, and external obliques play an active role. Specifically, the transversus abdominis, like the diaphragm, increases intra-abdominal pressure and supports trunk stabilization. However, the relationship between respiratory muscle strength and the endurance of core stability muscles remains unclear.

In light of this information, this study aims to investigate the relationship between the endurance of core muscles, which contribute to trunk stabilization, and respiratory parameters in children with thoracic hyperkyphosis.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 7 and 18
* Have a thoracic kyphosis angle (Cobb) of ≥45˚ on a lateral X-ray or a kyphosis index of ≤13

Exclusion Criteria:

* Individuals who have undergone major surgery or trauma related to the musculoskeletal system, particularly the spine and upper extremities
* Difficulty in understanding given instructions
* Presence of rigid deformity in the spine (Scheuermann's Kyphosis)
* Presence of congenital deformities (Congenital Kyphosis)

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: hildren with thoracic hyperkyphosis.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity | 2 weeks
  Forced vital capacity is the volume of gas expelled from the lungs in a fast, forced and deep expiration after a deep, forced inspiration. Forced vital capacity will be performed in a sitting position using a portable spirometer (Spirobank; MIR, Rome, Italy) according to American Thoracic Society guidelines.
Forced expiratory volume in the first second | 2 weeks
  Forced expiratory volume in the first second is the amount of air expelled from the lungs in the first second with forced expiration. Forced expiratory volume in the first second will be performed in a sitting position using a portable spirometer (Spirobank; MIR, Rome, Italy) according to American Thoracic Society guidelines.
Forced vital capacity/Forced expiratory volume Ratio | 2 weeks
  The Forced vital capacity/Forced expiratory volume Ratio, also called the modified Tiffeneau-Pinelli index, is a calculated ratio used in the diagnosis of obstructive and restrictive lung disease. The ratio will be performed in a sitting position using a portable spirometer (Spirobank; MIR, Rome, Italy) according to American Thoracic Society guidelines.
Peak expiratory flow rat | 2 weeks
  Peak expiratory flow rate is the volume of air forcefully expelled from the lungs in one quick exhalation, and is a reliable indicator of ventilation adequacy as well as airflow obstruction. The ratio will be performed in a sitting position using a portable spirometer (Spirobank; MIR, Rome, Italy) according to American Thoracic Society guidelines.
Respiratory Muscle Strength | 2 weeks
  Respiratory muscle strength will be assessed using maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) with an electronic pressure transducer
side bridge test | 2 weeks
  In the side bridge test, participants will begin in a side-lying position on their dominant side. When ready, they will be instructed to lift their hips without any verbal cues, supporting themselves with one arm. They will be asked to maintain a straight body line and hold this position for as long as possible. Participants will be instructed to place their free hand on their opposite shoulder. The duration for which they can maintain the position will be recorded in seconds.
prone bridge test | 2 weeks
  In the prone bridge test, participants will start in a prone position, supported on their knees and forearms. When they feel ready, they will be instructed to lift their knees off the ground without any verbal cues, maintaining a position supported by their forearms and toes. The duration for which they can hold this position will be recorded in seconds.
flexor endurance test | 2 weeks
  In the flexor endurance test, participants will begin in a supine position. When they feel ready, they will be instructed to pull their knees towards their chest in parallel with the ground without any verbal cues. They will then raise their upper body, lifting the lower edge of their scapula off the ground. The duration for which they can hold this position will be recorded in seconds.
Sorenson test | 2weeks
  In the Sorenson test, participants will start in a prone position on a stretcher, with their upper body resting on the stretcher. They will be repositioned so that the part of their body in contact with the bed is the anterior superior iliac spine. Participants will be instructed to hold onto the sides of a chair with their hands to maintain balance. A researcher will secure their legs, and when participants feel ready, they will cross both hands over their shoulders without any verbal instructions. They will be asked to hold the position parallel to the ground. The duration for which they can maintain this position will be recorded in seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided